CLINICAL TRIAL: NCT06514742
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Aticaprant 10 mg as Adjunctive Therapy in Adult Participants With Major Depressive Disorder (MDD) With Moderate-to-severe Anhedonia and Inadequate Response to Current Antidepressant Therapy and an Open Label Long-term Extension Treatment With Aticaprant
Brief Title: A Study of Aticaprant 10 mg as Adjunctive Therapy in Adult Participants With Major Depressive Disorder (MDD) With Moderate-to-severe Anhedonia and Inadequate Response to Current Antidepressant Therapy and Long-term Extension Treatment With Aticaprant
Acronym: VENTURA-7
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Early study termination due to insufficient efficacy.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 67953964MDD3007; 67953964MDD3007 (Other: Janssen Research & Development, LLC); 2024-511557-21-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Depressive Disorder, Major; Anhedonia
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aticaprant (Experimental)
  Interventions: Drug: Aticaprant
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aticaprant — Aticaprant tablet will be administered orally.
  Other Names: JNJ-67953964
  Arms: Aticaprant
Other: Placebo — Placebo tablet will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how well aticaprant works as compared with placebo when given along with an antidepressant therapy in improving the depressive symptoms in adult participants with major depressive disorder (MDD) with moderate to severe anhedonia (ANH+) who have not responded well to current antidepressant therapy with a selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI or SNRI).

ELIGIBILITY:
Inclusion Criteria:

* Be medically stable based on physical examination (including a brief neurologic examination), medical history, vital signs (including blood pressure), and 12-lead electrocardiogram (ECG) performed at screening and double blind (DB) baseline
* Meet diagnostic and statistical manual of mental disorders-5th edition (DSM-5) diagnostic criteria for recurrent or single episode major depressive disorder (MDD), without psychotic features (DSM-5 296.22, 296.23, 296.32, or 296.33), based upon clinical assessment and confirmed by the structured clinical interview for DSM-5 axis I disorders-clinical trials version (SCID-CT)
* Have symptoms of anhedonia based on clinical assessment and confirmed by presence of anhedonia (positive response to MDE module symptom Item 2) on the SCID-CT at screening
* Have had an inadequate response to at least 1 and up to 5 (inclusive) oral antidepressant treatments, administered at an adequate dose
* Is currently receiving and tolerating well any one of the following selective serotonin reuptake inhibitor or serotonin-norepinephrine reuptake inhibitor (SSRI or SNRI) antidepressants at screening, in any approved formulation and available in the participating country/territory: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, or desvenlafaxine at a stable dose (at or above the minimum therapeutic dose per Massachusetts general hospital antidepressant treatment response questionnaire (MGH ATRQ) for at least 6 weeks. The current antidepressant cannot be the first antidepressant treatment for the first lifetime episode of depression

Exclusion Criteria:

* Has had no response (treatment failure) to 2 or more consecutive antidepressant treatments administered at an adequate dose (at or above the minimum therapeutic dose) and duration (at least 6 weeks) in the current episode of depression including the current SSRI/SNRI (that is the one to be continued in the treatment phases) assessed using the MGH ATRQ
* Has one or more of the following diagnoses: (1) a current or prior (lifetime) DSM-5 diagnosis of: (a) a psychotic disorder or MDD with psychotic features, (b) bipolar or related disorders, (c) intellectual disability, (d) autism spectrum disorder, (e) borderline personality disorder, (f) antisocial personality disorder, (g) histrionic personality disorder, (h) narcissistic personality disorders, (i) somatoform disorders; (2) A primary DSM-5 diagnosis (which has been the primary focus of psychiatric treatment within the past 2 years) of: (a) panic disorder, (b) generalized anxiety disorder, (c) social anxiety disorder, (d) specific phobia; (3) A current (in the past year) DSM-5 diagnosis of: (a) obsessive-compulsive disorder, (b) post-traumatic stress disorder, (c) anorexia nervosa, (d) bulimia nervosa
* Has a history or evidence of clinically meaningful noncompliance with current antidepressant therapy
* Has a history of moderate-to-severe substance use disorder including alcohol use disorder according to DSM-5 criteria within 6 months before screening
* Has in the current depressive episode had vagal nerve stimulation or deep brain stimulation device in the current episode or has had an inadequate response to an adequate course of intravenous or intranasal ketamine or esketamine (greater than [>] 2 treatments), or electroconvulsive therapy (that is at least 7 treatments)
* Has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 3 months prior to the start of the screening phase, per the investigator's clinical judgment or based on the columbia suicidality severity rating scale (C-SSRS), corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) for suicidal ideation on the C-SSRS, or a history of suicidal behavior within the past 6 months prior to the start of the screening phase. Participants reporting suicidal ideation with intent to act or suicidal behavior at DB baseline should be excluded

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to Day 43 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score | Baseline to Day 43
  Change from baseline to Day 43 in MADRS total score will be reported.

SECONDARY OUTCOMES:
Change From Baseline to Day 43 in Dimensional Anhedonia Rating Scale (DARS) Total Score | Baseline to Day 43
  Change from baseline to Day 43 in DARS total score will be reported.
Change From Baseline to Day 43 in Changes in Sexual Function Questionnaire - 14 items (CSFQ-14) Total Score | Baseline to Day 43
  Change from baseline to Day 43 in CSFQ-14 total score will be reported.
Change From Baseline Over Time in MADRS Total Score | For double-blind (DB) treatment phase: Baseline (Day 1), Up to Day 43; For open-label (OL) treatment phase: Baseline (Day 43), Up to Week 31
  Change from baseline over time in the MADRS total score will be reported.
Percentage of responders on Depressive Symptoms Scale, Defined as a Greater Than or Equal to (>=) 50 Percent (%) Improvement in MADRS Total Score From Baseline to Day 43 | Baseline to Day 43
  Percentage of responders on depressive symptoms scale, defined as a >= 50 % improvement in MADRS total score from baseline to Day 43 will be reported.
Percentage of Participants With Remission of Depressive Symptoms, Defined as a MADRS Total Score Less Than or Equal to (<=)10 at Day 43 | Day 43
  Percentage of participants with remission of depressive symptoms, defined as a MADRS total score <=10 at Day 43 will be reported.
Change From Baseline to Day 43 in Patient Health Questionnaire, 9-item (PHQ-9) Total Score | Baseline to Day 43
  Change from baseline to Day 43 in the PHQ-9 total score will be reported.
Change From Baseline Over Time in DARS Total score. | For DB treatment phase: Baseline (Day 1), Up to Day 43; For OL treatment phase: Baseline (Day 43), Up to Week 31
  Change from baseline over time in DARS total score will be reported.
Change From Baseline Over Time in the PHQ-9 Anhedonia-Specific Item (PHQ-9, item 1). | For DB treatment phase: Baseline (Day 1), Up to Day 43; For OL treatment phase: Baseline (Day 43), Up to Week 31
  Change from baseline over time in the PHQ-9 Anhedonia-specific item (PHQ-9, Item 1) will be reported.
Percentage of Participants With a Score Less than (<) 2 in the PHQ-9 Anhedonia-specific Item (PHQ-9, Item 1) at Day 43 | Day 43
  Percentage of participants with a score < 2 in the PHQ-9 Anhedonia-specific Item (PHQ-9, Item 1) at Day 43 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (84):
- United States (39):
  - UAB Huntsville Regional Medical Campus, Huntsville, Alabama
  - IMA Clinical Research PC, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Advanced Research Center Inc, Anaheim, California
  - CI Trials, Bellflower, California
  - Behavioral Research Specialists LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - ATP Clinical Research, Orange, California
  - Lumos Clinical Research Center LLC, San Jose, California
  - Viking Clinical Research Ltd, Temecula, California
  - Sunwise Clinical Research, Walnut Creek, California
  - MCB Clinical Research Centers LLC, Colorado Springs, Colorado
  - Humanity Clinical Research Corp, Aventura, Florida
  - Elligo Independent Research Sites Mindful Behavioral Health, Boca Raton, Florida
  - Gulfcoast Medical Research Center, Fort Myers, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - LCC Medical Research Institute Inc, Miami, Florida
  - Floridian Clinical Research LLC, Miami, Florida
  - Medquest Translational Sciences, Miami Lakes, Florida
  - Best Choice Medical and Research Service, Pembroke Pines, Florida
  - K2 Medical Research, Tampa, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Accelerated Clinical Trials LLC, Peachtree Corners, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Fieve Clinical Research Inc, New York, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - OSU Department of Psychiatry and Behavioral Health, Columbus, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - UTHealth Houston Center for Interventional Psychiatry, Houston, Texas
  - Brain Health Consultants, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Perceptive Pharma Research, Richmond, Texas
  - Revival Research Institute LLC, Sherman, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Belgium (4):
  - Anima, Alken
  - Chu Tivoli, La Louvière
  - Centre Hospitalier Specialise Notre Dame Des Anges Asbl, Liège
  - Meclinas, Mechelen
- Brazil (4):
  - Universidade Federal do Ceara Hospital Universitario Walter Cantidio, Fortaleza
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - Centro Integrado Facili, São Bernardo do Campo
  - BR Trials, São Paulo
- Bulgaria (4):
  - Mental Health Center Prof. Dr. Ivan Temkov, Burgas
  - Medical Center Mentalcare OOD, Plovdiv
  - MHC - Sofia, EOOD, Sofia
  - Centre for Mental Health Prof.N.Shipkovenski EOOD, Sofia
- Finland (6):
  - Terveystalo Ruoholahti, Helsinki
  - Savon Psykiatripalvelu, Kuopio
  - Northern Clinical Trial Coordinators, Oulu
  - Oulu Mentalcare Oy, Oulu
  - Mehilainen Finlayson, Tampere
  - Clinical Research Services Turku - CRST, Turku
- Hungary (9):
  - Semmelweis Egyetem, Budapest
  - Eszak Budai Szent Janos Centrumkorhaz, Budapest
  - Processus Kft, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Gyor Moson Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Dr Mathe es Tarsa Bt, Kalocsa
  - Pte Aok Pszichiatriai Klinika, Pécs
  - PsychoTech Kft, Pécs
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
- Poland (5):
  - Osrodek Badan Klinicznych CLINSANTE S C Ewa Galczak Nowak Malgorzata Trzaska, Bydgoszcz
  - Centrum Zdrowia Alcea, Gdansk
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Osrodek Badan Klinicznych CLINSANTE S C, Torun
  - Ginemedica Sp. z o.o., Wroclaw
- Spain (8):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Institucion Hosp Hestia Palau, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Centro Salud Mental La Corredoria, Oviedo
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Prov. de Zamora, Zamora
- Sweden (5):
  - Affecta Pskyiatrimottagning, Halmstad
  - Linkoping University Hospital, Linköping
  - ProbarE i Lund AB, Lund
  - ProbarE i Stockholm AB, Stockholm
  - Studieenheten Akademiskt Specialistcentrum Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency